CLINICAL TRIAL: NCT04308681
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 2 Study of the Efficacy and the Safety and Tolerability of BMS-986278 in Participants With Pulmonary Fibrosis
Brief Title: A Study Measuring the Effectiveness, Safety, and Tolerability of BMS-986278 in Participants With Lung Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IM027-040; 2019-003992-21 (EudraCT Number)
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; Progressive Fibrotic Interstitial Lung Disease; Idiopathic interstitial pneumonia; Fibrotic interstitial pneumonia; Fibrotic interstitial lung disease; Fibrosing interstitial lung disease; Interstitial lung disease
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- IPF Dose 1 + Post Treatment Follow-up or OTE (Experimental): IPF (Idiopathic Pulmonary Fibrosis) OTE (Optional Treatment Extension)
  Interventions: Drug: BMS-986278
- IPF Dose 2 + Post Treatment Follow-up or OTE (Experimental)
  Interventions: Drug: BMS-986278
- IPF Placebo + Post Treatment Follow-up or OTE (Placebo Comparator)
  Interventions: Other: BMS-986278 Placebo
- PF-ILD Dose 1 + Post Treatment Follow-up or OTE (Experimental): PF-ILD (Progressive Fibrotic Interstitial Lung Disease)
  Interventions: Drug: BMS-986278
- PF-ILD Dose 2 + Post Treatment Follow-up or OTE (Experimental)
  Interventions: Drug: BMS-986278
- PF-ILD Placebo + Post Treatment Follow-up or OTE (Placebo Comparator)
  Interventions: Other: BMS-986278 Placebo

INTERVENTIONS:
Other: BMS-986278 Placebo — Specified Dose on Specified Days
  Arms: IPF Placebo + Post Treatment Follow-up or OTE; PF-ILD Placebo + Post Treatment Follow-up or OTE
Drug: BMS-986278 — Specified Dose on Specified Days
  Arms: IPF Dose 1 + Post Treatment Follow-up or OTE; IPF Dose 2 + Post Treatment Follow-up or OTE; PF-ILD Dose 1 + Post Treatment Follow-up or OTE; PF-ILD Dose 2 + Post Treatment Follow-up or OTE

SUMMARY:
The purpose of this study is to provide an initial evaluation of the effectiveness of BMS-986278 in participants with lung fibrosis, to demonstrate the safety of BMS-986278, and provide information on the drug levels of BMS-986278 in these participants.

ELIGIBILITY:
Inclusion Criteria:

For the idiopathic pulmonary fibrosis (IPF) Cohort

* Diagnosis of IPF within 7 years of screening
* Female and males ≥ 40 years of age

For the progressive fibrotic interstitial lung disease (PF-ILD) Cohort

* Evidence of progressive ILD within the 24 months before screening
* Female and male ≥ 21 years of age.

Exclusion Criteria:

* Women of childbearing potential (WOCBP)
* Active Smokers
* Current malignancy or previous malignancy up to 5 years prior to screening
* History of allergy to BMS-986278 or related compounds

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-08-04 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (118):
- United States (21):
  - Local Institution - 0032, Birmingham, Alabama
  - Local Institution, Phoenix, Arizona
  - Local Institution - 0028, Los Angeles, California
  - Local Institution - 0043, Stanford, California
  - University of Colorado Anschutz Medical Campus-Department of Medicine, Aurora, Colorado
  - Local Institution - 0006, Denver, Colorado
  - Local Institution - 0171, New Haven, Connecticut
  - Local Institution - 0035, Gainesville, Florida
  - Local Institution - 0166, Orlando, Florida
  - Local Institution - 0078, Atlanta, Georgia
  - Local Institution - 0031, Kansas City, Kansas
  - Local Institution - 0154, Baltimore, Maryland
  - Local Institution - 0003, Boston, Massachusetts
  - Local Institution - 0030, Chesterfield, Missouri
  - Local Institution - 0036, St Louis, Missouri
  - Local Institution - 0029, Cincinnati, Ohio
  - Local Institution - 0164, Columbus, Ohio
  - Local Institution, Hershey, Pennsylvania
  - Local Institution, Nashville, Tennessee
  - Local Institution - 0096, Charlottesville, Virginia
  - Local Institution, Falls Church, Virginia
- Argentina (6):
  - Local Institution - 0049, Buenos Aires, Distrito Federal
  - Local Institution - 0103, Rosario, Santa Fe Province
  - Local Institution - 0097, San Miguel de Tucumán, Tucumán Province
  - Local Institution - 0115, Buenos Aires
  - Local Institution - 0048, Buenos Aires
  - Local Institution - 0122, Mendoza
- Australia (8):
  - Local Institution - 0045, Camperdown, New South Wales
  - Local Institution - 0025, Westmead, New South Wales
  - Local Institution - 0026, Brisbane, Queensland
  - Local Institution - 0046, Greenslopes, Queensland
  - Local Institution - 0022, Adelaide, South Australia
  - Local Institution - 0023, Heidelberg, Victoria
  - Local Institution - 0021, Murdoch, Western Australia
  - Local Institution - 0044, Nedlands, Western Australia
- Belgium (3):
  - Local Institution - 0074, Brussels
  - Local Institution - 0065, Leuven
  - Local Institution - 0051, Liège
- Brazil (3):
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
  - Local Institution - 0076, São Paulo
- Canada (6):
  - Local Institution - 0141, Vancouver, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution - 0134, Toronto, Ontario
  - Local Institution - 0094, Montreal, Quebec
  - Local Institution - 0127, Québec, Quebec
  - Local Institution - 0144, Sherbrooke, Quebec
- Chile (3):
  - Local Institution - 0108, Curicó, Maule Region
  - Local Institution - 0054, Talca, Maule Region
  - Local Institution - 0038, Quillota, Región de Valparaíso
- China (4):
  - Local Institution - 0187, Beijing, Beijing Municipality
  - Local Institution - 0183, Beijing, Beijing Municipality
  - Local Institution - 0188, Wuhan, Hubei
  - Local Institution - 0189, Shanghai, Shanghai Municipality
- France (8):
  - Local Institution - 0120, Bobigny
  - Local Institution - 0066, Bron
  - Local Institution - 0136, Dijon
  - Local Institution - 0162, Marseille
  - Hopital Europeen Georges Pompidou, Paris
  - Local Institution - 0143, Paris
  - Local Institution - 0067, Rennes
  - Local Institution - 0132, Toulouse
- Germany (7):
  - Local Institution - 0111, Hanover, Lower Saxony
  - Local Institution - 0107, Essen
  - Local Institution, Freiburg im Breisgau
  - Local Institution - 0093, Großhansdorf
  - Local Institution - 0110, Heidelberg
  - Local Institution - 0121, Munich
  - Local Institution - 0119, Stuttgart
- Israel (5):
  - Local Institution - 0145, Tel Aviv, Tel Aviv
  - Local Institution - 0113, Haifa
  - Local Institution - 0149, Jerusalem
  - Local Institution - 0114, Petah Tikva
  - Local Institution - 0148, Ramat Gan
- Italy (4):
  - Local Institution - 0073, Catania
  - Local Institution - 0077, Modena
  - Local Institution - 0089, Monza
  - Local Institution - 0072, Roma
- Japan (16):
  - Local Institution - 0155, Seto, Aichi-ken
  - Local Institution - 0106, Kōriyama, Fukushima
  - Local Institution - 0180, Sapporo, Hokkaido
  - Local Institution - 0095, Kobe, Hyōgo
  - Local Institution - 0169, Kobe, Hyōgo
  - Local Institution - 0071, Yokohama, Kanagawa
  - Local Institution - 0112, Sakai, Osaka
  - Local Institution - 0128, Izumo, Shimane
  - Local Institution - 0064, Hamamatasu, Shizuoka
  - Local Institution - 0080, Bunkyo-ku, Tokyo
  - Local Institution - 0153, Minato-ku, Tokyo
  - Local Institution - 0177, Shinjyuku-ku, Tokyo
  - Local Institution - 0117, Kumamoto
  - Local Institution - 0146, Nagasaki
  - Local Institution - 0170, Saitama
  - Local Institution - 0173, Tokyo
- Mexico (5):
  - Local Institution, Mexico City, Mexico City
  - Local Institution - 0081, Monterrey, Nuevo León
  - Local Institution - 0109, Monterrey, N.l., Nuevo León
  - Local Institution - 0083, San Nicolás de los Garza, Nuevo León
  - Local Institution - 0156, Oaxaca City, Oaxaca
- South Korea (3):
  - Local Institution - 0087, Seoul
  - Local Institution - 0086, Seoul
  - Local Institution, Seoul
- Spain (8):
  - Local Institution, Barcelona
  - Local Institution - 0116, Barcelona
  - Local Institution - 0140, L'Hospitalet de Llobregat
  - Local Institution, Madrid
  - Local Institution - 0137, Madrid
  - Local Institution, Marbella Málaga
  - Local Institution - 0039, Pozuelo de Alarcón
  - Local Institution - 0147, Santander
- Taiwan (3):
  - Local Institution - 0176, Kaohsiung City
  - Local Institution - 0174, Taipei
  - Local Institution - 0175, Taipei
- United Kingdom (5):
  - Local Institution - 0050, Cambridge
  - Local Institution - 0163, Edinburgh
  - Local Institution - 0041, London
  - Local Institution - 0092, London
  - Local Institution, London

REFERENCES:
- [Derived] Kreuter M, Maher TM, Wuyts WA, Valenzuela C, Hamblin M, Kim S, Patel A, Elpers B, Richeldi L. Effect of Admilparant, a Lysophosphatidic Acid Receptor 1 Antagonist, on Disease Progression in Pulmonary Fibrosis. Chest. 2025 Sep;168(3):677-687. doi: 10.1016/j.chest.2025.04.003. Epub 2025 Apr 8. PMID 40210090
- [Derived] Corte TJ, Behr J, Cottin V, Glassberg MK, Kreuter M, Martinez FJ, Ogura T, Suda T, Wijsenbeek M, Berkowitz E, Elpers B, Kim S, Watanabe H, Fischer A, Maher TM. Efficacy and Safety of Admilparant, an LPA1 Antagonist, in Pulmonary Fibrosis: A Phase 2 Randomized Clinical Trial. Am J Respir Crit Care Med. 2025 Feb;211(2):230-238. doi: 10.1164/rccm.202405-0977OC. PMID 39393084
- [Derived] Corte TJ, Lancaster L, Swigris JJ, Maher TM, Goldin JG, Palmer SM, Suda T, Ogura T, Minnich A, Zhan X, Tirucherai GS, Elpers B, Xiao H, Watanabe H, Smith RA, Charles ED, Fischer A. Phase 2 trial design of BMS-986278, a lysophosphatidic acid receptor 1 (LPA1) antagonist, in patients with idiopathic pulmonary fibrosis (IPF) or progressive fibrotic interstitial lung disease (PF-ILD). BMJ Open Respir Res. 2021 Dec;8(1):e001026. doi: 10.1136/bmjresp-2021-001026. PMID 34969771
- [Derived] Cheng PTW, Kaltenbach RF 3rd, Zhang H, Shi J, Tao S, Li J, Kennedy LJ, Walker SJ, Shi Y, Wang Y, Dhanusu S, Reddigunta R, Kumaravel S, Jusuf S, Smith D, Krishnananthan S, Li J, Wang T, Heiry R, Sum CS, Kalinowski SS, Hung CP, Chu CH, Azzara AV, Ziegler M, Burns L, Zinker BA, Boehm S, Taylor J, Sapuppo J, Mosure K, Everlof G, Guarino V, Zhang L, Yang Y, Ruan Q, Xu C, Apedo A, Traeger SC, Cvijic ME, Lentz KA, Tirucherai G, Sivaraman L, Robl J, Ellsworth BA, Rosen G, Gordon DA, Soars MG, Gill M, Murphy BJ. Discovery of an Oxycyclohexyl Acid Lysophosphatidic Acid Receptor 1 (LPA1) Antagonist BMS-986278 for the Treatment of Pulmonary Fibrotic Diseases. J Med Chem. 2021 Nov 11;64(21):15549-15581. doi: 10.1021/acs.jmedchem.1c01256. Epub 2021 Oct 28. PMID 34709814
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who received 30 mg or 60 mg BMS-986278 in the 26-week long main study phase and met low BP criteria were given the option to receive 10 mg of BMS-986278 in the optional treatment extension (OTE), which lasted an additional 26 weeks.
  Participants who received placebo during the main study phase were re-randomized to receive either 30 mg or 60 mg of BMS-986278 in OTE.
  No participants received a 10 mg dose during the main study and no participants received placebo during the OTE.
Groups:
- IPF Cohort: Placebo: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort who received placebo twice a day for up to 26 weeks.
- IPF Cohort: 30 mg BMS-986278: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort received both 30 mg BMS-986278 and placebo twice per day for up to 26 weeks.
- IPF Cohort: 60 mg BMS-986278: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort received 60 mg BMS-986278 twice per day for up to 26 weeks.
- IPF Cohort - BMS-986278 10mg: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort who received 10 mg of BMS-986278 twice per day during the Optional Treatment Extension (OTE) phase only.
- PF-ILD Cohort: Placebo: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received placebo twice a day for up to 26 weeks.
- PF-ILD Cohort: 30 mg BMS-986278: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received both 30 mg BMS-986278 and placebo twice per day for up to 26 weeks.
- PF-ILD Cohort: 60 mg BMS-986278: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received both 60 mg BMS-986278 twice per day for up to 26 weeks.
- PF-ILD Cohort - 10mg BMS-986278: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received 10 mg of BMS-986278 during the Optional Treatment Extension (OTE) phase only. This arm includes participants who received 30 mg or 60 mg BMS-986278 BID in the main study who meet low BP criteria and were dose reduced to 10 mg BMS-986278 BID for the OTE.
Period: Pre-Treatment
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | IPF Cohort - BMS-986278 10mg | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278 | PF-ILD Cohort - 10mg BMS-986278
Started | 93 | 92 | 93 | 0 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Pre-Treatment Phase.) | 41 | 42 | 42 | 0 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Pre-Treatment Phase.)
Completed | 92 | 91 | 93 | 0 | 41 | 40 | 42 | 0
Not Completed | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Not reported | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Period: Treatment up to Week 26
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | IPF Cohort - BMS-986278 10mg | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278 | PF-ILD Cohort - 10mg BMS-986278
Started | 92 | 91 | 93 | 0 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Main Study.) | 41 | 40 | 42 | 0 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Main Study.)
Completed | 82 | 82 | 84 | 0 | 33 | 37 | 40 | 0
Not Completed | 10 | 9 | 9 | 0 | 8 | 3 | 2 | 0
Not completed — Withdrawal by participant | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Not completed — Other reasons | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Participant no longer meets study criteria | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 6 | 5 | 5 | 0 | 6 | 1 | 0 | 0
Not completed — Adverse event unrelated to study drug | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Period: OTE - 26 Weeks
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | IPF Cohort - BMS-986278 10mg | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278 | PF-ILD Cohort - 10mg BMS-986278
Started | 0 (Participants who received placebo in the Main Treatment phase were re-randomized to receive 30 mg or 60 mg BMS-986278 during the OTE.) | 100 | 102 | 11 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Main Study.) | 0 (Participants who received placebo in the Main Treatment phase were re-randomized to receive 30 mg or 60 mg BMS-986278 during the OTE.) | 41 | 46 | 4 (10 mg treatment was offered only in the OTE phase. No participants received 10 mg treatment during the Main Study.)
PBO BMS-986278 30 mg (Participants who received placebo treatment in the Main Study and received 30 mg of BMS-986278 in the Optional Treatment Extension (OTE) phase) | 0 | 33 | 0 | 0 | 0 | 13 | 0 | 0
PBO BMS-986278 60 mg (Participants who received placebo treatment in the Main Study and received 60 mg of BMS-986278 in the Optional Treatment Extension (OTE) phase) | 0 | 0 | 30 | 0 | 0 | 0 | 14 | 0
Completed | 0 | 96 | 89 | 8 | 0 | 39 | 42 | 4
Not Completed | 0 | 4 | 13 | 3 | 0 | 2 | 4 | 0
Not completed — Withdrawal by participant | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 8 | 3 | 0 | 1 | 2 | 0
Not completed — Adverse event unrelated to study drug | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics are reported for the safety population which is all treated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278 | Total
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42 | 399
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.0 (6.70) | 69.5 (7.31) | 68.8 (7.85) | 68.8 (8.06) | 71.4 (7.92) | 67.9 (8.41) | 69.5 (8.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 24 | 21 | 17 | 20 | 112
  Male | 76 | 77 | 69 | 20 | 23 | 22 | 287
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 18 | 19 | 7 | 6 | 9 | 80
  Not Hispanic or Latino | 39 | 36 | 37 | 19 | 21 | 22 | 174
  Unknown or Not Reported | 32 | 37 | 37 | 15 | 13 | 11 | 145
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 25 | 25 | 27 | 8 | 9 | 6 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 2 | 0 | 3
  White | 65 | 64 | 64 | 31 | 27 | 32 | 283
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 2 | 2 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (ppFVC) in IPF Participants
Description: Percent predicted forced vital capacity (ppFVC) is the percentage of predicted value per participant of forced vital capacity (FVC). FVC is defined as the maximum capacity of air that a participant can exhale after a maximum inspiration as measured by the volume of air exhaled in a spirometer. The data is reported as percent change from baseline in ppFVC. Percent change from baseline is a calculation that expresses the change in a value compared to its initial starting point (baseline) as a percentage, showing how much a value has increased or decreased relative to its original level; it's calculated by subtracting the baseline value from the new value, dividing by the baseline value, and then multiplying by 100%. The percent change in this endpoint was calculated from ppFVC values taken at baseline, which is defined as the measurement of ppFVC taken at first dose, and ppFVC values taken at Week 26. This endpoint reports data for the IPF cohort only as pre-specified in the protocol.
Time Frame: From baseline (first dose) up to week 26
Population: All treated participants in the IPF Cohort with baseline and week 26 results. Prespecified to be collected for IPF Cohort only.
Measure: Mean (Standard Error); unit: Percent change from baseline in ppFVC
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 70 | 59 | 67 | 0 | 0 | 0
Percent change from baseline in ppFVC | -2.807 (0.7286) | -3.068 (0.7335) | -1.120 (0.6691) |  |  |

2. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose up to 30 days after last dose during the main study treatment phase
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 74 | 69 | 69 | 32 | 33 | 28

3. Secondary Outcome: The Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose up to 30 days after last dose during the main study treatment phase
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 16 | 10 | 10 | 13 | 4 | 6

4. Secondary Outcome: The Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: The number of participants who discontinued study treatment due to adverse events (AEs)
Time Frame: From first dose up to 30 days after last dose during the main study treatment phase
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 9 | 9 | 6 | 7 | 1 | 0

5. Secondary Outcome: The Number of Participants Who Died Due to Adverse Events (AEs)
Description: The number of participants who died while receiving study treatment due to an adverse event
Time Frame: From first dose up to 30 days after last dose during the main study treatment phase
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 2 | 3 | 4 | 3 | 0 | 0

6. Secondary Outcome: Maximum Concentration (Cmax)
Description: Cmax is defined as the maximum concentration of the analyte recorded in the participants. Cmax of BMS-986278 and BMT-327319 was derived from plasma concentration versus time data.
Time Frame: On Day 1 and Week 4 (Day 29)
Population: All randomized participants who received at least one administration of BMS-986278 and had quantifiable concentration data
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 0 | 8 | 13 | 0 | 2 | 2
ng/mL
  Day 1; Analyte: BMS-986278: number analyzed (Participants) | 0 | 7 | 13 | 0 | 2 | 2
  Day 1; Analyte: BMS-986278 |  | 465.0 (36.23) | 1089.8 (42.06) |  | 715.4 (2.87) | 1112.3 (77.45)
  Day 1; Analyte: BMT-323719: number analyzed (Participants) | 0 | 7 | 13 | 0 | 2 | 2
  Day 1; Analyte: BMT-323719 |  | 114.66 (32.147) | 167.35 (39.538) |  | 94.8 (10.39) | 189.6 (86.07)
  Day 29; Analyte: BMS-986278 |  | 641.0 (27.68) | 1301.3 (20.80) |  | 691.9 (2.04) | 1247.80 (29.84)
  Day 29; Analyte: BMT-323719 |  | 169.30 (28.104) | 275.82 (34.554) |  | 161.9 (30.60) | 433.5 (58.73)

7. Secondary Outcome: Time to Maximum Concentration (Tmax)
Description: Tmax is defined as the amount of time until the maximum concentration of the analyte is recorded in the participants
Time Frame: On Day 1 and Week 4 (Day 29)
Population: as for outcome 6
Measure: Median (Full Range); unit: Hours
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 0 | 8 | 13 | 0 | 2 | 2
Hours
  Day 1; Analyte: BMS-986278: number analyzed (Participants) | 0 | 7 | 13 | 0 | 2 | 2
  Day 1; Analyte: BMS-986278 |  | 2.0170 [1.567 to 4.100] | 1.6670 [1.283 to 5.917] |  | 1.55 [1.50 to 1.60] | 2.01 [1.83 to 2.18]
  Day 1; Analyte: BMT-323719: number analyzed (Participants) | 0 | 7 | 13 | 0 | 2 | 2
  Day 1; Analyte: BMT-323719 |  | 4.0670 [1.867 to 7.900] | 4.0330 [1.900 to 8.000] |  | 7.96 [7.92 to 8.00] | 4.10 [3.98 to 4.22]
  Day 29; Analyte: BMS-986278: number analyzed (Participants) | 0 | 8 | 12 | 0 | 2 | 2
  Day 29; Analyte: BMS-986278 |  | 1.9080 [1.450 to 4.117] | 1.6750 [1.317 to 4.000] |  | 2.68 [1.533 to 3.82] | 4.06 [3.98 to 4.13]
  Day 29; Analyte: BMT-323719: number analyzed (Participants) | 0 | 8 | 12 | 0 | 2 | 2
  Day 29; Analyte: BMT-323719 |  | 4.0670 [2.083 to 6.000] | 2.0085 [1.417 to 7.850] |  | 5.79 [4.10 to 7.48] | 3.74 [1.48 to 6.00]

8. Secondary Outcome: Area Under Curve (AUC0-8)
Description: Area under the plasma concentration-time curve (AUC) from the timepoint of 0 hours to 24 hours post dose as measured on Day 1 and Week 4.
Time Frame: On Day 1 and Week 4 (Day 29)
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 0 | 7 | 12 | 0 | 2 | 2
h*ng/mL
  Day 1; Analyte: BMS-986278: number analyzed (Participants) | 0 | 6 | 9 | 0 | 2 | 2
  Day 1; Analyte: BMS-986278 |  | 1990.4530 (20.78185) | 4430.5891 (31.16188) |  | 3358 (8.7) | 4347 (61.3)
  Day 1; Analyte: BMT-323719: number analyzed (Participants) | 0 | 5 | 6 | 0 | 2 | 2
  Day 1; Analyte: BMT-323719 |  | 686.2045 (32.95587) | 913.4300 (50.72949) |  | 532 (NA) — Geometric coefficient of variation not calculated due to insufficient number of events | 2081 (NA) — Geometric coefficient of variation not calculated due to insufficient number of events
  Day 29; Analyte: BMS-986278 |  | 2853.9081 (21.72108) | 5433.1662 (25.62819) |  | 3591 (NA) — Geometric coefficient of variation not calculated due to insufficient number of events | 8107 (NA) — Geometric coefficient of variation not calculated due to insufficient number of events
  Day 29; Analyte: BMT-323719: number analyzed (Participants) | 0 | 4 | 8 | 0 | 0 | 2
  Day 29; Analyte: BMT-323719 |  | 1179.6486 (31.27987) | 1784.7369 (30.32795) |  |  | 2839 (45.8)

9. Secondary Outcome: Concentration Trough (Ctrough)
Description: Ctrough is defined as the lowerst concentration of drug in the blood immediately before the next dose is administered
Time Frame: On Week 4 (Day 29) and Week 12 (Day 85)
Population: as for outcome 6
Measure: Median (Full Range); unit: ng/mL
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 0 | 56 | 60 | 0 | 28 | 31
ng/mL
  Day 29-BMS-986278: number analyzed (Participants) | 0 | 51 | 48 | 0 | 24 | 31
  Day 29-BMS-986278 |  | 92.1 [13.5 to 433] | 217 [32.4 to 1540] |  | 116.0000 [26.300 to 392.000] | 286.0000 [49.600 to 2659.000]
  Day 85-BMS-986278 |  | 84.2 [16.7 to 389] | 199 [5.37 to 726] |  | 88.7000 [20.100 to 380.000] | 196.0000 [68.000 to 1773.000]
  Day 29-BMT-323719: number analyzed (Participants) | 0 | 49 | 47 | 0 | 24 | 30
  Day 29-BMT-323719 |  | 60.3 [12.9 to 207] | 141 [52.4 to 384] |  | 75.5000 [0.200 to 121.000] | 177.5000 [0.200 to 693.000]
  Day 85-BMT-323719 |  | 64.2 [0.200 to 174] | 132 [0.200 to 371] |  | 67.4500 [11.000 to 186.000] | 156.0000 [0.200 to 326.000]

10. Secondary Outcome: The Number of Participants Experiencing Electrocardiogram (ECG) Abnormalities
Description: A frequency summary of investigator clinical interpretation of ECG abnormal findings is listed.
Time Frame: At Week 26
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 27 | 18 | 31 | 5 | 9 | 12

11. Secondary Outcome: Change From Baseline in Vital Sign Measurements
Description: The change from baseline in select vital sign measurements. Baseline is defined as first dose.
Time Frame: At baseline and Week 26
Population: All treated participants with baseline and week 26 vital sign measurement results.
Measure: Median (Full Range); unit: Change from baseline in mmHg
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 77 | 72 | 79 | 27 | 33 | 37
Change from baseline in mmHg
  Sitting Diastolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 77 | 71 | 79 | 27 | 33 | 37
  Sitting Diastolic Blood Pressure - 0 Hours Pre-Dose | 0.0 [-20 to 19] | 0.0 [-21 to 20] | 1.0 [-16 to 24] | 3.0 [-9 to 13] | 1.0 [-18 to 17] | -1.0 [-27 to 15]
  Standing Diastolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 71 | 72 | 77 | 26 | 32 | 37
  Standing Diastolic Blood Pressure - 0 Hours Pre-Dose | -2.0 [-18 to 15] | 0.0 [-28 to 22] | 1.0 [-24 to 30] | 1.5 [-15 to 26] | -0.5 [-14 to 20] | 0.0 [-18 to 16]
  Supine Diastolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 73 | 72 | 78 | 26 | 33 | 37
  Supine Diastolic Blood Pressure - 0 Hours Pre-Dose | -1.0 [-12 to 18] | 1.0 [-25 to 17] | 1.0 [-23 to 19] | 2.5 [-13 to 15] | 0.0 [-8 to 17] | 0.0 [-14 to 14]
  Sitting Systolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 77 | 71 | 79 | 27 | 33 | 37
  Sitting Systolic Blood Pressure - 0 Hours Pre-Dose | -1.0 [-29 to 37] | 1.0 [-23 to 30] | 3.0 [-22 to 34] | 0.0 [-35 to 17] | 1.0 [-22 to 37] | -1.0 [-49 to 34]
  Standing Systolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 71 | 72 | 77 | 26 | 32 | 37
  Standing Systolic Blood Pressure - 0 Hours Pre-Dose | -3.0 [-27 to 28] | -1.5 [-35 to 31] | 3.0 [-28 to 36] | 0.5 [-38 to 33] | 0.5 [-23 to 28] | 0.0 [-34 to 26]
  Supine Systolic Blood Pressure - 0 Hours Pre-Dose: number analyzed (Participants) | 73 | 72 | 78 | 26 | 33 | 37
  Supine Systolic Blood Pressure - 0 Hours Pre-Dose | 0.0 [-24 to 34] | 0.0 [-25 to 43] | 3.0 [-24 to 24] | 2.5 [-29 to 25] | 2.0 [-20 to 49] | -3.0 [-30 to 23]

12. Secondary Outcome: Change From Baseline in Percent Predicted Forced Vital Capacity (ppFVC) in PF-ILD Participants
Description: Percent predicted forced vital capacity (ppFVC) is the percentage of predicted value per participant of forced vital capacity (FVC). FVC is defined as the maximum capacity of air that a participant can exhale after a maximum inspiration as measured by the volume of air exhaled in a spirometer. The data is reported as percent change from baseline in ppFVC. Percent change from baseline is a calculation that expresses the change in a value compared to its initial starting point (baseline) as a percentage, showing how much a value has increased or decreased relative to its original level; it's calculated by subtracting the baseline value from the new value, dividing by the baseline value, and then multiplying by 100%. The percent change in this endpoint was calculated from ppFVC values taken at baseline, which is defined as the measurement of ppFVC taken at first dose, and ppFVC values taken at Week 26. This endpoint reports data for PF-ILD cohort only as pre-specified in the protocol.
Time Frame: At baseline and Week 26
Population: All treated participants in the PF-ILD Cohort with baseline and week 26 results. Pre-specified to be collected for PF-ILD Cohort only.
Measure: Mean (Standard Error); unit: Percent change from baseline
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 0 | 0 | 0 | 22 | 29 | 31
Percent change from baseline |  |  |  | -2.681 (1.4730) | 2.717 (0.9054) | -1.203 (0.8808)

13. Secondary Outcome: The Number of Participants With ≥ 10% Absolute Decline in ppFVC (%)
Description: The number of participants with ≥ 10% absolute decline in percent predicted forced vital capacity (ppFVC) at pre-specified timepoints.
  ppFVC is the maximum capacity of air that a participant can exhale after a maximum inspiration. It measures the volume of air exhaled in a spirometer, after a maximal inspiration. It is reported as the percentage of the predicted value for the participant.
  The number of participants represented signify the number of participants with applicable data during the specific visit at the specific timepoint.
Time Frame: At Weeks 4, 8, 12, 16, 20, and 26
Population: All treated participants with ppFVC data during visits at the specific time windows of Weeks 4, 8, 12, 16, 20, and 26.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 78 | 75 | 75 | 35 | 30 | 36
Participants
  Week 4 | 3 | 0 | 2 | 0 | 0 | 0
  Week 8: number analyzed (Participants) | 77 | 72 | 69 | 34 | 30 | 34
  Week 8 | 4 | 4 | 3 | 2 | 0 | 0
  Week 12: number analyzed (Participants) | 76 | 69 | 74 | 32 | 27 | 34
  Week 12 | 4 | 1 | 3 | 1 | 0 | 0
  Week 16: number analyzed (Participants) | 78 | 71 | 71 | 30 | 29 | 34
  Week 16 | 3 | 2 | 2 | 2 | 0 | 0
  Week 20: number analyzed (Participants) | 75 | 60 | 66 | 28 | 27 | 31
  Week 20 | 10 | 1 | 1 | 2 | 1 | 0
  Week 26: number analyzed (Participants) | 70 | 59 | 67 | 22 | 29 | 31
  Week 26 | 7 | 7 | 4 | 3 | 3 | 1

14. Secondary Outcome: The Number of Participants With 0% Change in ppFVC (%)
Description: The number of participants with 0% change in percent predicted forced vital capacity (ppFVC) at pre-specified timepoints.
  ppFVC is the maximum capacity of air that a participant can exhale after a maximum inspiration. It measures the volume of air exhaled in a spirometer, after a maximal inspiration. It is reported as the percentage of the predicted value for the participant.
Time Frame: Weeks 4, 8, 12, 16, 20, and 26
Population: All treated participants with ppFVC data at the prespecified timepoints Weeks 4, 8, 12, 16, 20, and 26.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 78 | 75 | 75 | 35 | 30 | 36
Participants
  Week 4 | 48 | 41 | 33 | 14 | 12 | 13
  Week 8: number analyzed (Participants) | 77 | 72 | 69 | 34 | 30 | 34
  Week 8 | 47 | 43 | 69 | 15 | 13 | 12
  Week 12: number analyzed (Participants) | 76 | 69 | 74 | 32 | 27 | 34
  Week 12 | 46 | 43 | 39 | 17 | 13 | 13
  Week 16: number analyzed (Participants) | 78 | 71 | 71 | 30 | 29 | 34
  Week 16 | 51 | 45 | 39 | 15 | 11 | 18
  Week 20: number analyzed (Participants) | 75 | 60 | 66 | 28 | 27 | 31
  Week 20 | 51 | 40 | 33 | 18 | 15 | 18
  Week 26: number analyzed (Participants) | 70 | 59 | 67 | 22 | 29 | 31
  Week 26 | 53 | 42 | 34 | 17 | 22 | 19

15. Secondary Outcome: Time to First Occurrence ≥ 10% Absolute Decline in ppFVC (%)
Description: The amount of time in weeks to the participant's first occurrence ≥ 10% absolute decline in Percent Predicted Forced Vital Capacity (ppFVC). A participant's time is censored at the last observed time prior to discontinuation if a participant discontinues study without event, or at week 26 if a participant does not experience the event until the end of week 26. Kaplan-Meier product limit method will be employed to estimate the survival curves.
  ppFVC is the maximum capacity of air that a participant can exhale after a maximum inspiration. It measures the volume of air exhaled in a spirometer, after a maximal inspiration. It is reported as the percentage of the predicted value for the participant.
Time Frame: From first dose up to the first occurrence of ≥ 10% absolute decline in ppFVC
Population: The total accumulated number of participants with ≥ 10% Absolute Decline in ppFVC events at any time from first dose up to Week 26. A participant's time was censored at the last observed time prior to discontinuation if a participant discontinues study without event, or at week 26 if a participant does not experience the event until the end of week 26.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 16 | 9 | 6 | 5 | 5 | 1
Weeks | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower and upper limit not calculated due to insufficient number of events. | NA [26.3 to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events.

16. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Forced Vital Capacity (ppFVC)
Description: The absolute change in ppFVC (%) is measured from baseline up to the pre-specified timepoints of Weeks 4, 8, 12, 16, 20, and 26.
  ppFVC is the maximum capacity of air that a participant can exhale after a maximum inspiration. It measures the volume of air (mL) exhaled in a spirometer, after a maximal inspiration. It is reported as the percentage of the predicted value for the participant.
Time Frame: From baseline up to Weeks 4, 8, 12, 16, 20, and 26
Population: All treated participants with ppFVC data at Weeks 4, 8, 12, 16, 20, and 26
Measure: Mean (Standard Deviation); unit: Percentage of predicted value
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 78 | 75 | 75 | 35 | 30 | 36
Percentage of predicted value
  Absolute change from Baseline to Week 4 | -1.491 (4.3773) | -0.482 (4.2499) | 0.023 (5.4007) | 1.119 (6.0123) | 0.327 (3.1862) | 0.217 (3.5946)
  Absolute change from Baseline to Week 8: number analyzed (Participants) | 77 | 72 | 69 | 34 | 30 | 34
  Absolute change from Baseline to Week 8 | -1.783 (4.5234) | -1.046 (4.8192) | -1.079 (5.1294) | -0.334 (7.6326) | 0.966 (3.2631) | 0.475 (3.2802)
  Absolute change from Baseline to Week 12: number analyzed (Participants) | 76 | 69 | 74 | 32 | 27 | 34
  Absolute change from Baseline to Week 12 | -1.974 (5.0324) | -0.589 (4.8575) | -1.109 (5.9152) | -2.012 (5.5436) | 0.114 (4.2490) | 0.196 (3.7168)
  Absolute change from Baseline to Week 16: number analyzed (Participants) | 78 | 71 | 71 | 30 | 29 | 34
  Absolute change from Baseline to Week 16 | -2.422 (5.0040) | -1.042 (5.1644) | -1.220 (4.3475) | -1.180 (7.6897) | -0.197 (4.5490) | -0.394 (4.3439)
  Absolute change from Baseline to Week 20: number analyzed (Participants) | 75 | 60 | 66 | 28 | 27 | 31
  Absolute change from Baseline to Week 20 | -2.625 (4.8978) | -1.717 (3.9049) | -0.387 (4.2802) | -2.650 (4.2813) | -0.382 (4.6328) | -0.272 (6.0198)
  Absolute change from Baseline to Week 26: number analyzed (Participants) | 70 | 59 | 67 | 22 | 29 | 31
  Absolute change from Baseline to Week 26 | -2.807 (6.0959) | -3.068 (5.6339) | -1.120 (5.4768) | -2.681 (6.9089) | -2.717 (4.8758) | -1.203 (4.9043)

17. Secondary Outcome: Absolute Change From Baseline in Forced Vital Capacity (FVC)
Description: Forced vital capacity (FVC) is defined as the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible. The absolute change in FVC (mL) is measured from baseline up to Weeks 4, 8, 12, 16, 20, and 26.
Time Frame: From baseline up to Weeks 4, 8, 12, 16, 20, and 26
Population: All treated participants with FVC data at Weeks 4, 8, 12, 16, 20, and 26
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 78 | 75 | 75 | 35 | 30 | 36
mL
  Absolute change from Baseline to Week 4 | -54.7 (153.50) | -21.2 (142.25) | 4.3 (181.75) | 39.1 (152.57) | 6.0 (107.11) | -0.30 (113.07)
  Absolute change from Baseline to Week 8: number analyzed (Participants) | 77 | 72 | 69 | 34 | 30 | 34
  Absolute change from Baseline to Week 8 | -62.7 (157.81) | -38.2 (173.96) | -36.1 (165.74) | -8.8 (180.10) | 24.7 (92.87) | 11.2 (106.11)
  Absolute change from Baseline to Week 12: number analyzed (Participants) | 76 | 69 | 74 | 32 | 27 | 34
  Absolute change from Baseline to Week 12 | -75.5 (184.02) | -27.2 (173.23) | -35.4 (176.48) | -61.6 (177.42) | -1.5 (129.64) | 0.9 (128.40)
  Absolute change from Baseline to Week 16: number analyzed (Participants) | 78 | 71 | 71 | 30 | 29 | 34
  Absolute change from Baseline to Week 16 | -88.2 (183.44) | -41.0 (184.89) | -45.8 (152.79) | -44.3 (222.44) | -22.8 (146.75) | -12.1 (140.79)
  Absolute change from Baseline to Week 20: number analyzed (Participants) | 75 | 60 | 66 | 28 | 27 | 31
  Absolute change from Baseline to Week 20 | -95.6 (181.41) | -70.0 (142.70) | -21.1 (154.05) | -84.6 (134.01) | -15.2 (168.21) | -3.9 (222.29)
  Absolute change from Baseline to Week 26: number analyzed (Participants) | 70 | 59 | 67 | 22 | 29 | 31
  Absolute change from Baseline to Week 26 | -106.4 (214.94) | -117.3 (207.60) | -48.8 (184.97) | -99.1 (212.04) | -100.0 (166.30) | -37.7 (179.38)

18. Secondary Outcome: Absolute Change From Baseline in Single Breath Diffusing Capacity of Carbon Monoxide (DLCO SB)
Description: The absolute change in single breath diffusing capacity of carbon monoxide (DLCO SB) (mL/min/mmHg) (corrected for hemoglobin) from baseline to Week 26. DLCO is defined as a measurement of the extent to which oxygen passes from the alveoli into the blood. Baseline is defined as first dose.
Time Frame: From baseline up to Week 26
Population: All treated participants with DLCO SB data at Week 26
Measure: Median (Full Range); unit: mL/min/mmHg
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 43 | 40 | 44 | 20 | 32 | 32
mL/min/mmHg | -0.4664 [-17.023 to 5.725] | -0.3418 [-14.024 to 3.190] | -0.4518 [-5.449 to 3.888] | -0.2352 [-15.031 to 9.564] | -0.3269 [-8.902 to 2.086] | -0.1829 [-12.766 to 7.063]

19. Secondary Outcome: Absolute Change From Baseline in Percent Predicted Single Breath Diffusing Capacity of Carbon Monoxide (ppDLCO SB)
Description: The absolute change in percent predicted single breath diffusing capacity of carbon monoxide (DLCO SB) (mL/min/mmHg) (corrected for hemoglobin) from baseline to Week 26. DLCO is defined as a measurement of the extent to which oxygen passes from the alveoli into the blood. Baseline is defined as first dose.
Time Frame: From baseline up to Week 26
Population: All treated participants with ppDLCO SB data at Week 26
Measure: Median (Full Range); unit: Percentage of predicted value
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 44 | 40 | 44 | 21 | 33 | 34
Percentage of predicted value | -1.4634 [-38.133 to 64.451] | -0.3470 [-26.548 to 51.300] | -3.2455 [-48.939 to 35.463] | -1.000 [-22.176 to 11.587] | -1.4683 [-62.971 to 13.767] | -1.4609 [-13.016 to 20.997]

20. Secondary Outcome: Absolute Change From Baseline in Walking Endurance/Distance
Description: The absolute change in walking endurance/distance as determined by the 6-minute walk test (6MWT) from baseline to Week 26. The 6-Minute Walk Test (6MWT) is a submaximal exercise test used to assess aerobic capacity and endurance. Baseline is defined as first dose.
Time Frame: From baseline up to Week 26
Population: All participants with evaluable 6MWT data at Week 26
Measure: Median (Full Range); unit: Meters
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 67 | 62 | 70 | 25 | 33 | 37
Meters | 0.0 [-495 to 119] | 3.0 [-260 to 138] | 6.0 [-370 to 92] | 11.0000 [-315.833 to 175.000] | 0.0000 [-220.000 to 188.400] | -14.0000 [-173.000 to 242.857]

21. Secondary Outcome: Time to First Acute Exacerbation
Description: Time to first acute exacerbations of lung fibrosis was measured from the day of first dose up to the day of first acute exacerbation. Participants who discontinued the study treatment prior to the end of the main study without experiencing the event were excluded from the analysis. A participant's time was censored at the last observed time prior to discontinuation if a participant discontinued study without event, or at week 26 if a participant did not experience the event until the end of week 26.
  Acute exacerbations were defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality, as follows:
  1. Acute worsening or development of dyspnea (< 1 month duration)
  2. Imaging with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia
  3. Respiratory deterioration not fully explained by cardiac failure or fluid overload
Time Frame: From the first dose up to the day of the first acute exacerbation or Week 26, whichever comes first
Population: All participants who experienced acute exacerbation
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 2 | 3 | 1 | 3 | 0 | 1
Weeks | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events. |  | NA [NA to NA] — Median, lower limit, and upper limit not calculated due to insufficient number of events.

22. Secondary Outcome: The Number of Participants Experiencing Acute Exacerbation
Description: The number of participants experiencing acute exacerbations of lung fibrosis.
  Acute exacerbations were defined as an acute, clinically significant, respiratory deterioration characterized by evidence of new widespread alveolar abnormality, as follows:
  1. Acute worsening or development of dyspnea (< 1 month duration)
  2. Imaging with new bilateral ground-glass opacity and/or consolidation superimposed on a background pattern consistent with usual interstitial pneumonia
  3. Respiratory deterioration not fully explained by cardiac failure or fluid overload
Time Frame: From the first dose up to the day of the first acute exacerbation or Week 26, whichever comes first
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Cohort: Placebo | IPF Cohort: 30 mg BMS-986278 | IPF Cohort: 60 mg BMS-986278 | PF-ILD Cohort: Placebo | PF-ILD Cohort: 30 mg BMS-986278 | PF-ILD Cohort: 60 mg BMS-986278
Number analyzed (Participants) | 92 | 91 | 93 | 41 | 40 | 42
Participants | 2 | 3 | 1 | 3 | 0 | 1

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 58 weeks). SAEs and Other AEs were assessed from first dose to 30 days following last dose (up to approximately 58 weeks).
Groups:
- IPF Cohort - Main Study - Placebo: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort who received placebo twice a day for up to 26 weeks.
- IPF Cohort - Main Study - 30 mg BMS-986278: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort received both 30 mg BMS-986278 and placebo twice per day for up to 26 weeks.
- IPF Cohort - Main Study - BMS-986278 60mg: Participants in the Progressive Fibrotic Idiopathic Pulmonary Fibrosis (IPF) cohort received 60 mg BMS-986278 twice per day for up to 26 weeks.
- IPF Cohort - OTE Phase - PBO BMS-986278 30 mg; PF-ILD Cohort - OTE Phase - PBO BMS-986278 30mg: Participants who received placebo treatment in the Main Study and received 30 mg of BMS-986278 in the Optional Treatment Extension (OTE)
- IPF Cohort - OTE Phase - PBO BMS-986278 60mg; PF-ILD Cohort - OTE Phase - PBO BMS-986278 60mg: Participants who received placebo treatment in the Main Study and received 60 mg of BMS-986278 in the Optional Treatment Extension (OTE)
- PF-ILD Cohort - Main Study - Placebo: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received placebo twice a day for up to 26 weeks.
- PF-ILD Cohort - Main Study - BMS-986278 30mg: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received both 30 mg BMS-986278 and placebo twice per day for up to 26 weeks.
- PF-ILD Cohort - Main Study - BMS-986278 60mg: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received 60 mg BMS-986278 twice per day for up to 26 weeks.
- PF-ILD Cohort - OTE Phase - BMS-986278 10mg: Participants in the Progressive Fibrotic Interstitial Lung Disease (PF-ILD) cohort who received 10 mg of BMS-986278 during the Optional Treatment Extension (OTE) phase only.
Arm/Group | IPF Cohort - Main Study - Placebo | IPF Cohort - Main Study - 30 mg BMS-986278 | IPF Cohort - Main Study - BMS-986278 60mg | IPF Cohort - BMS-986278 10mg | IPF Cohort - OTE Phase - PBO BMS-986278 30 mg | IPF Cohort - OTE Phase - PBO BMS-986278 60mg | PF-ILD Cohort - Main Study - Placebo | PF-ILD Cohort - Main Study - BMS-986278 30mg | PF-ILD Cohort - Main Study - BMS-986278 60mg | PF-ILD Cohort - OTE Phase - BMS-986278 10mg | PF-ILD Cohort - OTE Phase - PBO BMS-986278 30mg | PF-ILD Cohort - OTE Phase - PBO BMS-986278 60mg
All-Cause Mortality (participants affected / at risk) | 4/92 | 4/91 | 5/93 | 3/11 | 4/100 | 6/102 | 4/41 | 0/40 | 0/42 | 0/4 | 1/41 | 3/46
Serious Adverse Events (participants affected / at risk) | 16/92 | 10/91 | 10/93 | 4/11 | 19/100 | 23/102 | 13/41 | 4/40 | 6/42 | 0/4 | 8/41 | 7/46
Other Adverse Events (participants affected / at risk) | 57/92 | 54/91 | 51/93 | 8/11 | 40/100 | 43/102 | 19/41 | 23/40 | 24/42 | 4/4 | 18/41 | 23/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Cohort - Main Study - Placebo (N=92) | IPF Cohort - Main Study - 30 mg BMS-986278 (N=91) | IPF Cohort - Main Study - BMS-986278 60mg (N=93) | IPF Cohort - BMS-986278 10mg (N=11) | IPF Cohort - OTE Phase - PBO BMS-986278 30 mg (N=100) | IPF Cohort - OTE Phase - PBO BMS-986278 60mg (N=102) | PF-ILD Cohort - Main Study - Placebo (N=41) | PF-ILD Cohort - Main Study - BMS-986278 30mg (N=40) | PF-ILD Cohort - Main Study - BMS-986278 60mg (N=42) | PF-ILD Cohort - OTE Phase - BMS-986278 10mg (N=4) | PF-ILD Cohort - OTE Phase - PBO BMS-986278 30mg (N=41) | PF-ILD Cohort - OTE Phase - PBO BMS-986278 60mg (N=46)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1
Pneumonia legionella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Forced vital capacity decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Lung squamous cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatic nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal dermatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Idiopathic interstitial pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 0 | 1 | 8 | 7 | 1 | 0 | 0 | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IPF Cohort - Main Study - Placebo (N=92) | IPF Cohort - Main Study - 30 mg BMS-986278 (N=91) | IPF Cohort - Main Study - BMS-986278 60mg (N=93) | IPF Cohort - BMS-986278 10mg (N=11) | IPF Cohort - OTE Phase - PBO BMS-986278 30 mg (N=100) | IPF Cohort - OTE Phase - PBO BMS-986278 60mg (N=102) | PF-ILD Cohort - Main Study - Placebo (N=41) | PF-ILD Cohort - Main Study - BMS-986278 30mg (N=40) | PF-ILD Cohort - Main Study - BMS-986278 60mg (N=42) | PF-ILD Cohort - OTE Phase - BMS-986278 10mg (N=4) | PF-ILD Cohort - OTE Phase - PBO BMS-986278 30mg (N=41) | PF-ILD Cohort - OTE Phase - PBO BMS-986278 60mg (N=46)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Constipation (Gastrointestinal disorders) | 5 | 0 | 5 | 1 | 2 | 2 | 1 | 1 | 2 | 0 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 10 | 11 | 1 | 4 | 8 | 6 | 6 | 3 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 3 | 5 | 4 | 0 | 1 | 0 | 3 | 4 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Fatigue (General disorders) | 4 | 5 | 1 | 0 | 2 | 4 | 1 | 0 | 3 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 4 | 1 | 1 | 4 | 5 | 2 | 1 | 0 | 1 | 2 | 3
COVID-19 (Infections and infestations) | 7 | 3 | 9 | 1 | 12 | 8 | 2 | 5 | 6 | 1 | 7 | 6
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 6 | 3 | 0 | 3 | 1 | 0 | 1 | 3 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 3 | 1 | 0 | 3 | 1 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 0 | 3 | 0 | 1 | 0 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 4 | 3 | 1 | 1 | 3 | 1 | 0 | 2 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 2 | 0 | 1 | 1 | 4 | 0 | 4 | 0 | 0 | 2
Dizziness exertional (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 6 | 5 | 0 | 3 | 4 | 3 | 1 | 2 | 0 | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 10 | 1 | 3 | 7 | 4 | 3 | 5 | 1 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 4 | 0 | 3 | 6 | 6 | 2 | 0 | 0 | 2 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 1 | 3 | 6 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 3 | 7 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 2 | 4 | 1 | 0 | 3 | 0 | 4 | 3 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 9 | 7 | 5 | 1 | 3 | 0 | 1 | 2 | 4 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/81/NCT04308681/Prot_SAP_000.pdf